CLINICAL TRIAL: NCT04972708
Title: Genetics of COVID-19 Risks & Resilience in Bipolar Disorder as Subproject of BIPGEN (Genetic Changes in Bipolar Disorder)
Brief Title: Genetics of COVID-19 Risks & Resilience in Bipolar Disorder
Acronym: BIPCOVID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 23-199 ex 10/11
Record Dates: First submitted 2021-07-21; First posted 2021-07-22 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Bipolar Disorder; Covid19; Stress
Keywords: bipolar disorder; covid-19 pandemic
MeSH Terms: conditions — Bipolar Disorder; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA from blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bipolar Disorder: 100 patients after COVID-19 infection 100 patients without COVID-19 infection
  Interventions: Genetic: Cross-sectional genetics study
- Healthy controls: 100 controls after COVID-19 infection 100 controls without COVID-19 infection
  Interventions: Genetic: Cross-sectional genetics study

INTERVENTIONS:
Genetic: Cross-sectional genetics study — Cross-sectional genetics study

SUMMARY:
BIPGEN is a cross-sectional study on the genetics of bipolar disorder. As a subproject of BIPGEN, BIP-COVID is a cross-sectional genetics study about risks & resilience in the COVID-19 (Coronavirus disease) pandemic in bipolar disorder (BD) and healthy controls at the Medical University of Graz. Study participants with BD and controls from the well-established BIPLONG and BIPGEN studies will undergo a special BIP-COVID visit, which will include a COVID-19 specific online Lime survey about the psychological burden in the COVID-19 crisis, a COVID-19 antibody test (IgM and IgG), inflammation markers and isolation of DNA from fasting blood. Genotyping of DNA will be done with the GSA V.3 array. Genetic analyses (Polygenic Risk Scores of I. Stress or Major Depression and II. COVID-19 infection established with the programs PLINK, PRSice and R) will be used to analyze the genetic mechanisms of COVID-19 pandemic associated psychological symptoms and COVID-19 infection risk. Systems biology methods will be used to depict protective pathways against COVID-19 infection (e.g. Lithium pathways) and against COVID-19 associated psychiatric symptoms.

DETAILED DESCRIPTION:
Methods: BIPGEN is a cross-sectional study on the genetics of bipolar disorder (BD). BIPGEN includes a personality questionnaire (TEMPS-A). DNA is isolated in the BIPGEN study from fasting blood with the QUIASYMPHONY robot from study participants with Bipolar Disorder (diagnosis according to DSM-IV) and healthy controls. The DNA is then genotyped with classic genotyping arrays (GWAS array). The aim of BIPGEN is to associate genetic variants (single-nucleotide-polymorphisms/ SNPs or copy-number-variations/CNVs) with bipolar affective disorder.

A subproject of BIPGEN is the BIP-COVID project, which is a cross-sectional genetics study about risks & resilience in the COVID-19 pandemic in BD and healthy controls at the Medical University of Graz. Study participants with BD and controls from the well-established BIPLONG and BIPGEN studies will undergo a special BIP-COVID visit, which will include a COVID-19 specific online Lime survey about the psychological burden in the COVID-19 crisis, a COVID-19 antibody test (IgM and IgG), inflammation markers and isolation of DNA from fasting blood. Genotyping of DNA will be done with the GSA V.3 array. Genetic analyses (Polygenic Risk Scores of I. Stress or Major Depression and II. COVID-19 infection established with the programs PLINK, PRSice and R) will be used to analyze the genetic mechanisms of COVID-19 pandemic associated psychological symptoms and COVID-19 infection risk. Systems biology methods will be used to depict protective pathways against COVID-19 infection (e.g. Lithium pathways) and against COVID-19 associated psychiatric symptoms

Aim:

1. We aim at analyzing the neuropsychological and genetic underpinning of COVID-19 associatedreactive psychiatric symptoms in BD and in healthy controls.
2. We aim at analyzing genetic predictors of COVID-19 infection in BD and in controls.
3. We aim at analyzing the protective effects of the GSK-3β inhibitor lithium against COVID-19 infection.

Intervention: Cross-sectional genetics study

Key inclusion and exclusion criteria: Inclusion criteria are written consent after previous written and verbal information, diagnosis of BD according to DSM-IV and age between 18 and 75 years. Exclusion criteria include acute suicidality, lack of consent, severe active drug dependence (i.e., alcohol, benzodiazepines, morphine), other currently active severe mental / cerebral organic disease (e.g. epilepsy, brain tumor), severe skull-brain trauma / brain surgery in the past, known florid tumor disease, congenital / infantile mental retardation, dementia (from Mini-Mental State Examination (MMSE) 20), severe florid autoimmune diseases or current immunosuppression (e.g., lupus erythematosus, HIV (human immunodeficiency virus), multiple sclerosis), cardiac, renal and pulmonary disorders or PTSD (post-traumatic stress disorder) or anxiety.

Healthy controls do not have a history of mental disorder and do not have first- or second-degree relatives with psychiatric disorders.

Primary and secondary endpoint(s) of the BIPCOVID project:

The primary endpoint is PRS of stress, the secondary endpoint is PRS of COVID-19 risk.

Sample size, statistical analyses, power calculation: The program G*Power (Version 3.1) was used for the calculation of the number of cases. Linear bivariate regression analyses for two groups (BD and control cohort) will be calculated with the results from psychological/psychiatric inventories as predictors (e.g. Pittsburgh Sleep Quality Index, Mediterranean Diet Score, Resilience Scale) and the three PRS as criterion. G*Power calculates for a linear bivariate regression, with a Δ slope of 0.03, α = .05 and a power of 95 % a total sample size of 364 persons.

Trial duration of BIPCOVID: 3 years.

Participating centers: The BIP-COVID sample will be recruited as monocentric study at the special outpatient department for Bipolar Disorders (managed by Univ.Prof. Eva Reininghaus) at the Department of Psychiatry and Psychotherapeutic Medicine at the Medical University of Graz, Austria. Psychiatric genetics and bioinformatics experts from the University of Basel, the University of Marburg, the University of Bonn, the Karolinska Institutet & Medical University of Vienna & CAMH Toronto will supervise the KLIF-funded doctoral student and will support the state-of-the-art bioinformatics analyses.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria are written consent after previous written and verbal information, diagnosis of BD according to DSM-IV and age between 18 and 75 years.

Exclusion Criteria:

Exclusion criteria include

* acute suicidality
* lack of consent
* severe active drug dependence (i.e., alcohol, benzodiazepines, morphine)
* other currently active severe mental / cerebral organic disease (e.g. epilepsy, brain tumor),
* severe skull-brain trauma / brain surgery in the past,
* known florid tumor disease,
* congenital / infantile mental retardation,
* dementia (from MMSE 20),
* severe florid autoimmune diseases or current immunosuppression (e.g., lupus erythematosus, HIV, multiple sclerosis),
* cardiac, renal and pulmonary disorders or PTSD or anxiety
* Healthy controls do not have a history of mental disorder and do not have first- or second-degree relatives with psychiatric disorders.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants with bipolar disorder and healty controls
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
PRS of stress or depression | 3 Years
  genetic sum score for depression (polygenic risk score)- the higher the score, the higher the risk
PRS of COVID-19 infection | 3 Years
  genetic sum score for COVID-19 infection (polygenic risk score)- the higher the score, the higher the risk

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No